CLINICAL TRIAL: NCT06547658
Title: The Heterogeneous Effects of Mouth Closure on Airflow in Patients With Obstructive Sleep Apnea
Brief Title: The Effect of Mouth Closure on Airflow in OSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Massachusetts Eye and Ear Infirmary (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, David Andrew Wellman, Professor, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2019P002847; R01HL128658 (NIH)
Record Dates: First submitted 2024-08-01; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Hypopnea, Sleep
Keywords: Obstructive sleep apnea; Mouth breathing; Upper airway; Drug-induced sleep endoscopy
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Mouth Breathing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mouth closed (Experimental): Closing the mouth by applying pressure to the mentum until the teeth were in occlusion, without altering the head position. Performed during flow-limited breathing.
  Interventions: Other: Mouth closure
- Mouth relaxed (No Intervention): Mouth in the natural relaxed position during sleep.

INTERVENTIONS:
Other: Mouth closure — Closing the mouth during sleep by applying pressure to the mentum until the teeth were in occlusion, without altering the head position.
  Arms: Mouth closed

SUMMARY:
Mouth breathing is associated with increased airway resistance, pharyngeal collapsibility, and obstructive sleep apnea (OSA) severity. It is commonly believed that closing the mouth can mitigate the negative effects of mouth breathing during sleep. However, we propose that mouth breathing serves as an essential route bypassing obstruction along the nasal route (e.g., velopharynx). The present study investigates the role of mouth breathing as an essential route in some OSA patients and its association with upper airway anatomical factors.

Participants underwent drug-induced sleep endoscopy (DISE) with simultaneous pneumotach airflow measurements through the nose and mouth separately. During the DISE procedure, alternating mouth closure (every other breath) cycles were performed during flow-limited breathing.

We evaluated the overall effect mouth closure on inspiratory airflow, and the change in inspiratory airflow with mouth closure across three mouth-breathing quantiles. We also evaluated if velopharyngeal obstruction was associated with mouth breathing and a negative airflow response to mouth closure.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed obstructive sleep apnea (AHI > 5 events/h).
* Scheduled to undergo clinical drug-induced sleep endoscopy.

Exclusion Criteria:

* pregnancy
* age under 18 years
* poor general health
* allergy to propofol or dexmedetomidine
* history of surgical treatment for sleep apnea, such as palate, tongue base, or epiglottis surgery.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-12-17 (Actual); Primary Completion 2022-07-10 (Actual); Study Completion 2022-07-10 (Actual)

PRIMARY OUTCOMES:
Total inspiratory flow | 1 day - the intervention of mouth closure on the outcome is applied acutely on alternating breaths, such that the effect of mouth closure is assessed based on the experiment which occurs in a single day.
  Change in airflow in the transition from mouth relaxed to mouth closed (intervention).

SECONDARY OUTCOMES:
Change in total inspiratory airflow with mouth closure | 1 day - the intervention of mouth closure is applied acutely on alternating breaths, such that the effect of mouth closure on the outcome is assessed based on the experiment which occurs in a single day.
  We analyzed the change in total inspiratory flow within three quantiles of roughly equal sample sizes based on oral breathing; quantile 1: oral airflow <0.05 L/min, quantile 2: oral airflow between 0.05 and 2.2 L/min, and quantile 3: oral airflow >2.2 L/min.
  We also analyzed the effect of velopharyngeal obstruction on the change in total inspiratory airflow.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to make the IPD available to other researchers.

REFERENCES:
- [Derived] Yang H, Huyett P, Wang TY, Sumner J, Azarbarzin A, Labarca GPT, Messineo L, Gell LK, Aishah A, Hu WH, White DP, Sands SA, Wellman A, Vena D. Mouth Closure and Airflow in Patients With Obstructive Sleep Apnea: A Nonrandomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2024 Nov 1;150(11):1012-1019. doi: 10.1001/jamaoto.2024.3319. PMID 39361293